CLINICAL TRIAL: NCT01466244
Title: PTEN Determination in Squamous Cell Cancer of The Head and Neck Treated on E5397, A Randomized Phase III Trial of Cisplatin Plus Placebo Versus Cisplatin Plus C225 (Cetuximab) in Metastatic/Recurrent Head and Neck Cancer
Brief Title: Biomarkers in Patients With Metastatic or Recurrent Head and Neck Cancer Treated With Cisplatin and Cetuximab on ECOG-E5397
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000715505; ECOG-E5397T3
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Cancer
Keywords: metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IVA squamous cell carcinoma of the larynx; stage IVA squamous cell carcinoma of the lip and oral cavity; stage IVA squamous cell carcinoma of the oropharynx; stage IVA squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IVB squamous cell carcinoma of the larynx; stage IVB squamous cell carcinoma of the lip and oral cavity; stage IVB squamous cell carcinoma of the oropharynx; stage IVB squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IVC squamous cell carcinoma of the larynx; stage IVC squamous cell carcinoma of the lip and oral cavity; stage IVC squamous cell carcinoma of the oropharynx; stage IVC squamous cell carcinoma of the paranasal sinus and nasal cavity; untreated metastatic squamous neck cancer with occult primary
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Cisplatin; Gene Expression Profiling; Microarray Analysis; Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Biological: cetuximab
Drug: cisplatin
Genetic: gene expression analysis
Genetic: microarray analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is studying biomarkers in patients with metastatic or recurrent head and neck cancer treated with cisplatin and cetuximab on ECOG-E5397.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare cetuximab activity, as reflected in response rate (RR), in PTEN-deficient and PTEN-expressing cancers.

Secondary

* Examine RR, progression-free survival (PFS), and overall survival (OS) in PTEN-deficient and PTEN-expressing cancers, by treatment arm.

OUTLINE: Tissue microarray slides collected earlier from ECOG-E5397 are immunostained with PTEN antibody and analyzed with AQUA.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Treated on protocol ECOG-E5397

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients enrolled on E5397 from who samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2011-11-11 (Actual); Primary Completion 2012-01-11 (Actual); Study Completion 2012-01-11 (Actual)

PRIMARY OUTCOMES:
Cetuximab activity as reflected in RR | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Burtness, MD, Principal Investigator — Fox Chase Cancer Center